CLINICAL TRIAL: NCT04983836
Title: Comparison of Analgesic Efficiency Between Serratus Block and Paravertebral Block in Video-assisted Thoracic Surgery. Double-blind Randomized Comparative Non-inferiority Study
Brief Title: Comparison of Analgesic Efficiency Between Serratus Block and Paravertebral Block in Video-assisted Thoracic Surgery. Double-blind Randomized Comparative Non-inferiority Study (BSBP)
Acronym: BSBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 19-AOI-04
Record Dates: First submitted 2021-07-19; First posted 2021-07-30 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: Prospective, comparative, monocentric, randomized non-inferiority interventional study, in double-blind.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Block (Experimental)
  Interventions: Procedure: Serratus anesthesia technique
- Paravertebral Block (Other)
  Interventions: Procedure: Paravertebral anesthesia technique

INTERVENTIONS:
Procedure: Serratus anesthesia technique — locoregional anaesthesia allowing analgesia of the hemi-thorax by ultrasound guided single injection of naropeine 5mg/ml
  Arms: Serratus Block
Procedure: Paravertebral anesthesia technique — Ultrasound guided single injection of of naropeine 5mg/ml dose into the paravertebral space next to the thoracic spine
  Arms: Paravertebral Block

SUMMARY:
Currently, the 2 main techniques of regional loco anesthesia in perioperative analgesic management of the thoracotomy remains the establishment of a thoracic epidural or paravertebral block. On the other hand, there is no standard of perioperative analgesic management in the case of thoracic surgery under video-thoracoscopy. The video-thoracoscopy, by its mini-invasive character, makes the levels of pain lower in post-operative questioning the benefit/risk balance of the paravertebral block. In 2013, Blanco published a new technique of locoregional anesthesia called the block Serratus allowing analgesia of a homolateral thorax hemi The latter by its simplicity of realization and its lesser risk is growing in thoracic surgery. This pilot study finds an equivalence in total oxycodone consumption in the first 2 post-operative days with a number of complications related to the serratus block lower than the serratus block compared to the paravertebral block in preoperative surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient who has given their free, informed and signed consent
* Social security affiliation;

Exclusion Criteria:

* pregnant woman
* guardianship / curatorship / private patient under public law
* surgery to be performed urgently (less than 24 hours)
* surgery redux
* thoracotomy surgery
* sternotomy surgery
* pleurectomy
* patient participating simultaneously in another research that may interfere with results of the study
* severe abnormality of haemostasis (80,000/ml platelets) and/or coagulation (TP 50%, factor V 50%).
* Prior use of morphine;
* chronic pain/chest neuropathies
* sepsis
* patients with insulin-dependent diabetes and/or diabetic neuropathy.
* severe kidney or liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-12-05 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Pain evaluation | 48 hours after the surgery
  Assess the non-inferiority of the single-injection echo-guided serratus block, performed in video-thoracic surgery preoperative, on the post-operative mean pain during the first 48 hours, compared to the single-injection echo-guided paravertebral block with a simple numeric scale (from 0 to 10)

SECONDARY OUTCOMES:
Walking test | 24 hours after the surgery
  Improvement of walking distance during the test at 6 min post-operative
Post operative morphine dose Post operative administrated morphin dose | 48 hours after the surgery
  Mesure of intraoperative morphine administrated dose and total morphine administrated dose (in mg).
Morphine side effect quantification | 48 hours after the surgery
  Collection of adverse reactions due to morphine administration (nausea, vomiting, pruritus, urine retention, respiratory depression)
Length of hospitalisation duration | 1 year
  Number of hospitalisation days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, Toutes, France

IPD SHARING:
Plan to Share IPD: No
No data sharing in planned